CLINICAL TRIAL: NCT02809222
Title: Kinetics of the Plasmatic Concentration of L-Ascorbic Acid in Patient With Myelodysplastic Syndromes and Control Subjects
Brief Title: Plasmatic L-AScorbic Acid in MYelodyplastic Syndroms and Controls
Acronym: PLASMYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Tours Autogreffe (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PHAO16-EG/PLASMYC; 2016-A00539-42 (Registry Identifier: IdRCB)
Record Dates: First submitted 2016-06-17; First posted 2016-06-22 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Myelodysplastic Syndrome; Secondary Acute Myeloid Leukemia
Keywords: Myelodysplastic syndrome; Ascorbic acid; Oxidative stress; Preleukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Preleukemia | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with MDS at diagnosis (Other): The intervention, specific to the study, is to take blood samples on patients with MDS at diagnosis. A quality of life questionnaire will also be used to monitor patients
  Interventions: Other: Samples; Other: Quality of life questionnaire
- Patients with MDS in treatment (Other): The intervention, specific to the study, is to take blood samples on patients with MDS receiving treatment. A quality of life questionnaire will also be used to monitor patients
  Interventions: Other: Samples; Other: Quality of life questionnaire
- Healthy volunteers (Other): The intervention, specific to the study, is to take blood samples on patients healthy volunteers.
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — Blood samples
Other: Quality of life questionnaire — Questionnaire to assess the quality of life of cancer patients
  Other Names: EORTC QLQ-C30
  Arms: Patients with MDS at diagnosis; Patients with MDS in treatment

SUMMARY:
Myelodysplastic syndromes (MDS) is a group of heterogeneous diseases characterised by the clonal evolution of dysplastic hematopoietic stem cells. This evolution is associated with accumulation of cytogenetic mutations which leads to acute myeloid leukaemia (AML). Evolution of MDS is also associated with increase of reactive oxygen species (ROS). The increase of ROS is associated with accumulation of cytogenetic mutations. Ascorbic acid (AA) is an actor of the regulation of the oxidative metabolism in the human body.

Studies showed that supplementation with AA can change the proliferation status of MDS cells. Adjuvant treatment with AA is associated with a beneficial effect on the evolution of MDS and AML. The present study aim at describing the variations of plasmatic ascorbic acid concentrations between healthy volunteers and patients with myelodysplastic syndromes advanced in their treatment or recently diagnosed during a follow-up of 12 months.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) is a group of heterogeneous life threatening diseases characterised by the clonal evolution of dysplastic myeloid hematopoietic stem cells. This evolution is initially associated with an excess of apoptosis followed by an excess of proliferation then, after accumulation of cytogenetic mutations, a transformation in acute myeloid leukaemia (AML) can appear. Evolution of MDS is also associated with increase of reactive oxygen species (ROS) . In MDS mice, perturbations of the metabolism of ROS is associated with increases in the number of cytogenetic mutations.

Ascorbic acid (AA) is an actor of the regulation of the oxidative metabolism in the human body. In vitro studies showed that supplementation with AA can change the proliferation status of MDS cells . Guinea pigs with a phenotype with excess of ROS supplemented with AA have less somatic mutations and less MDS. Adjuvant treatment with AA is associated with a beneficial effect on the evolution of MDS and AML.

To our knowledge no study have demonstrated the variations of the parameters of the oxidative metabolism during the evolution of MDS. The present study aim at describing the variations of plasmatic ascorbic acid concentrations between healthy volunteers and patients diagnosed with MDS in treatment or recently diagnosed during a follow-up of 12 months. During the follow-up a collection of plasma from volunteers and patients will be created for later analysis.

ELIGIBILITY:
1. Patients MDS "at diagnosis" group selection criteria

   Inclusion Criteria:
   * Diagnosis of myelodysplastic syndrome according to the 2008 WHO classification
   * Patient diagnosed for less than 4 months before inclusion
   * Patient untreated by other means than blood transfusions
   * Age ≥ 60 years
   * Patient affiliated to social security scheme
   * Informed consent signed by the patient

   Exclusion Criteria:
   * Previous allogenic stem cell transplantation
   * Patient with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
   * Active inflammatory disease
   * Patient under legal protection measure
   * Patient unwilling or who cannot submit to prospective biological follow-up
2. Patients MDS "in treatment" group selection criteria:

   Inclusion Criteria:
   * Diagnosis of myelodysplastic syndrome according to the 2008 WHO classification
   * Patient not included in patients MDS "at diagnosis" group
   * Patient diagnosed for more than 12 months
   * Treated with hypomethylating agents and/or erythropoiesis-stimulating agents and/or blood transfusions.
   * Age ≥ 60 years
   * Patient affiliated to social security scheme
   * Informed consent signed by the patient

   Exclusion Criteria:
   * Previous allogenic stem cell transplantation
   * Patient with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
   * Active inflammatory disease
   * Patient under legal protection measure
   * Patient unwilling or who cannot submit to prospective biological follow-up
3. Healthy volunteers group selection criteria:

Inclusion Criteria:

* Age ≥ 60 years
* Patient affiliated to social security scheme
* Informed consent signed by the patient

Exclusion Criteria:

* History of another primary malignancy that is currently clinically significant or currently requires active intervention
* History of active inflammatory diseases
* Volunteer under legal protection measure
* Volunteer unwilling or who cannot submit to prospective biological follow-up

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Plasmatic ascorbic acid concentration at baseline | month 0
  For all groups: Plasmatic ascorbic acid concentration at first visit (0 month)

SECONDARY OUTCOMES:
Plasmatic ascorbic acid concentration during follow-up | at 3 months, 6 months and 12 months
  For all groups: Plasmatic ascorbic acid concentrations at 6 months and 12 months visits with an extra plasmatic ascorbic acid concentrations at 3 months for patients MDS groups
Plasmatic antioxidants concentrations | at 0 months, 6 months and 12 months
  For all groups: Plasmatic antioxidants concentrations at 0 months, 6 months and 12 months
Collection of plasma | at 0 month, 3 months, 6 months and 12 months
  For all groups: Creation of a collection of plasma samples for later analysis at 0 month, 6 months and 12 months with an extra plasma sample at 3 months for patients MDS groups
Complete blood count and blood blasts cells | at 0 month, 3 months, 6 months and 12 months
  For patients MDS groups: Complete blood count and blood blasts cells at 0 month, 3 months, 6 months and 12 months
Polyunsaturated fatty acids | at 0 month, 3 months, 6 months and 12 months
  For patients MDS groups: Polyunsaturated fatty acids at 0 month, 3 months, 6 months and 12 months
Plasmatic ascorbic acid concentration and number of adverse events | at 3 months, 6 months and 12 months
  For patients MDS groups: Plasmatic ascorbic acid concentration at 3 months, 6 months and 12 months and number of adverse events during follow-up
Oxidative stress parameters and number of adverse events | at 3 months, 6 months and 12 months
  For patients MDS groups: Oxidative stress parameters at 3 months, 6 months and 12 months and number of adverse events during follow-up
Plasmatic ascorbic acid concentration and parameters of iron metabolism | at 0 month and 12 months
  For patients MDS groups: Plasmatic ascorbic acid concentration and parameters of iron metabolism at 0 month and 12 months
Plasmatic ascorbic acid concentration and quality of life | at 0 month, 3 months, 6 months and 12 months
  For patients MDS groups: Plasmatic ascorbic acid concentration and quality of life evaluated by the EORTC QLQ-C30 3rd version at 0 month, 3 months, 6 months and 12 months
Collection of frozen cells | 0 month and in case of evolution of the disease
  For patients MDS groups: Creation of a collection of frozen cells for DNA analysis at 0 month and in case of evolution of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel GYAN, MD,PhD, Principal Investigator — University Hospital, Tours
Locations (2):
- France (2):
  - Clinical Research Center, University Hospital, Tours, Tours
  - Department of Haematology and Cell Therapy, University Hospital, Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Das A, Dey N, Ghosh A, Das T, Chatterjee IB. NAD(P)H: quinone oxidoreductase 1 deficiency conjoint with marginal vitamin C deficiency causes cigarette smoke induced myelodysplastic syndromes. PLoS One. 2011;6(5):e20590. doi: 10.1371/journal.pone.0020590. Epub 2011 May 31. PMID 21655231
- [Background] Ghoti H, Amer J, Winder A, Rachmilewitz E, Fibach E. Oxidative stress in red blood cells, platelets and polymorphonuclear leukocytes from patients with myelodysplastic syndrome. Eur J Haematol. 2007 Dec;79(6):463-7. doi: 10.1111/j.1600-0609.2007.00972.x. Epub 2007 Nov 1. PMID 17976187
- [Background] Hole PS, Darley RL, Tonks A. Do reactive oxygen species play a role in myeloid leukemias? Blood. 2011 Jun 2;117(22):5816-26. doi: 10.1182/blood-2011-01-326025. Epub 2011 Mar 11. PMID 21398578
- [Background] Chung YJ, Robert C, Gough SM, Rassool FV, Aplan PD. Oxidative stress leads to increased mutation frequency in a murine model of myelodysplastic syndrome. Leuk Res. 2014 Jan;38(1):95-102. doi: 10.1016/j.leukres.2013.07.008. Epub 2013 Aug 16. PMID 23958061
- [Background] Levine M, Rumsey SC, Daruwala R, Park JB, Wang Y. Criteria and recommendations for vitamin C intake. JAMA. 1999 Apr 21;281(15):1415-23. doi: 10.1001/jama.281.15.1415. PMID 10217058
- [Background] Park CH. Vitamin C in leukemia and preleukemia cell growth. Prog Clin Biol Res. 1988;259:321-30. PMID 3362876
- [Background] Park CH, Kimler BF. Growth modulation of human leukemic, preleukemic, and myeloma progenitor cells by L-ascorbic acid. Am J Clin Nutr. 1991 Dec;54(6 Suppl):1241S-1246S. doi: 10.1093/ajcn/54.6.1241s. PMID 1962577
- [Background] Park CH, Kimler BF, Bodensteiner D, Lynch SR, Hassanein RS. In vitro growth modulation by L-ascorbic acid of colony-forming cells from bone marrow of patients with myelodysplastic syndromes. Cancer Res. 1992 Aug 15;52(16):4458-66. PMID 1643638
- [Background] Park CH, Kimler BF, Yi SY, Park SH, Kim K, Jung CW, Kim SH, Lee ER, Rha M, Kim S, Park MH, Lee SJ, Park HK, Lee MH, Yoon SS, Min YH, Kim BS, Kim JA, Kim WS. Depletion of L-ascorbic acid alternating with its supplementation in the treatment of patients with acute myeloid leukemia or myelodysplastic syndromes. Eur J Haematol. 2009 Aug;83(2):108-18. doi: 10.1111/j.1600-0609.2009.01252.x. Epub 2009 Mar 5. PMID 19284416
- [Background] Parker JE, Fishlock KL, Mijovic A, Czepulkowski B, Pagliuca A, Mufti GJ. 'Low-risk' myelodysplastic syndrome is associated with excessive apoptosis and an increased ratio of pro- versus anti-apoptotic bcl-2-related proteins. Br J Haematol. 1998 Dec;103(4):1075-82. doi: 10.1046/j.1365-2141.1998.01114.x. PMID 9886323
- [Background] Parker JE, Mufti GJ, Rasool F, Mijovic A, Devereux S, Pagliuca A. The role of apoptosis, proliferation, and the Bcl-2-related proteins in the myelodysplastic syndromes and acute myeloid leukemia secondary to MDS. Blood. 2000 Dec 1;96(12):3932-8. PMID 11090080
- [Background] Saito N, Miyamoto M, Gotoh U, Yoshitomi S. Effect of biscoclaurine alkaloids, prednisolone and ascorbic acid on myelodysplastic syndrome with pancytopenia: a case report. Eur J Haematol. 2000 Jan;64(1):61-5. doi: 10.1034/j.1600-0609.2000.9l036.x. No abstract available. PMID 10680708
- [Background] Welch JS, Klco JM, Gao F, Procknow E, Uy GL, Stockerl-Goldstein KE, Abboud CN, Westervelt P, DiPersio JF, Hassan A, Cashen AF, Vij R. Combination decitabine, arsenic trioxide, and ascorbic acid for the treatment of myelodysplastic syndrome and acute myeloid leukemia: a phase I study. Am J Hematol. 2011 Sep;86(9):796-800. doi: 10.1002/ajh.22092. Epub 2011 Aug 3. No abstract available. PMID 21815182